

### **Study Protocol**

## Lay Health Educators (LHEs)

LHEs will be invited to attend 2 training sessions (6 hours, orientation and intervention delivery) over Zoom. During the training sessions, our research team will provide LHEs Orientation Training Manual, which contains background information, project objectives, project description, LHE's responsibilities/activities, compensation/assistance, RCT participant's responsibilities/rights/activities, frequently asked questions, and handling challenging situations. LHEs will also receive the instruction to contact the research team if they do not know how to address the situation. The research team will ask LHEs to respect the privacy of others by keeping confidential any information they learn about others during meetings and calls.

#### Coordinators

Coordinators will not receive any training.

## **RCT** participants

All individuals recruited by the schools and teachers will receive an email from the research team that includes the consent information for the study and a link to the online baseline survey. They may choose to participate by themselves (individually) or participate with a family member who meets the eligibility criteria to participate together. We anticipate each school to recruit at least five individuals. Those who agree to participate in the study and complete the survey will be assigned to either the LHE condition or the control condition, depending on the group assignment of schools they are recruited from. Within the two weeks, after each participant completes the baseline survey, an OTC COVID-19 antigen test kit, which FDA authorizes under a EUA, will be provided to each participant. LHE participants will receive 1) LHE outreach/support (2 small group educational sessions via Zoom and 2 individual follow-up calls), 2) short video clips via email on the project overview and the guide to using a test kit (created by the research team in Korean and English), 3) test kits with written instructions on COVID-19 testing by Centers for Disease Control and Prevention (CDC) in English and Korean, and 4) weekly email reminders to report the use of COVID-19 at home antigen test kits. LHE outreach small group educational session is about 1 hour with 2 to 6 people. LHE will present COVID-19 testing and related information (including vaccination and safety practices).

Participants who participate as dyads (self-selected participation mode) are expected to attend the educational sessions together. At this educational session, LHE will provide education using PowerPoint presentations with easy-to-understand messages using culturally appropriate images and simple texts to present current information on 1) COVID-

19 testing; 2) relevance or reasons for getting tested; 3) the current guidelines for testing/ who should be tested; 4) types of tests available (e.g. PCR, antigens, and antibodies tests in the forms of nose swap and saliva tests); 5) understanding test results (positive versus negative) and the limitation of such tests (false negative); 6) the importance of repeated testing, discuss and address barriers for testing. LHE sessions provide a socially and culturally acceptable platform to engage participants to share personal stories, ask questions, and address concerns. At the end of each session, participants are encouraged to choose an "action item" from their 'Healthy Action Plan' to advance their knowledge and/or take steps toward making informed decisions about testing, and, if appropriate, taking steps toward getting tested. Participants have found that the LHE outreach session, follow-up call, and a 'Healthy Action Plan' have facilitated behavioral change by keeping them accountable. LHE may provide as-needed assistance to help a participant use a COVID-19 at-home antigen test kit, including demonstrating the use of the test kit.

# Statistical Analysis Plan

We will first conduct cross-sectional analyses of baseline data and compare baseline participant characteristics by groups/conditions. Differences in participant characteristics between groups will be included as covariates in subsequent analyses. We will use generalized linear mixed models using COVID-19 testing receipt based on self-report by participants as the outcome, with random effects for school, LHE, participant and family as needed to account for correlation within and between participants. We will then explore association between structural, sociocultural, and behavioral factors at individual, interpersonal, and community levels in association with COVID-19 testing receipt over time.